CLINICAL TRIAL: NCT05272865
Title: Pharmacokinetic and Pharmacodynamic Evaluation of 3 Standard Formulations of Δ9-THC in Healthy Volunteers and Post-chemotherapy Patients in Colombia
Brief Title: Pharmacokinetic and Pharmacodynamic Evaluation of Formulations of Δ9-THC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LaSanta S A S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1171735
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Nausea Post Chemotherapy; Vomiting; Cancer Pain; Cancer Related Pain; Neoplasms
Keywords: Dronabinol; THC; Cannabinoids; Cannabigerol; Cannabichromene; Pharmacokinetic and pharmacodynamic
MeSH Terms: conditions — Vomiting; Cancer Pain; Neoplasms | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dronabinol 5mg/mL (Active Comparator): Drug: Dronabinol (SYNDROS) Oral solution of SYNDROS (5 mg/mL)
  Interventions: Drug: Pharmacokinetic and pharmacodynamic profile of THC oral formulations with Dronabinol as comparator
- THC F1 (Experimental): Drug: THC Oral solution of THC (5 mg/mL)
  Interventions: Drug: Pharmacokinetic and pharmacodynamic profile of THC oral formulations with Dronabinol as comparator
- THC F2 (Experimental): Drug: THC:CBG Oral solution of THC (5 mg/mL) & CBG (5 mg/mL)
  Interventions: Drug: Pharmacokinetic and pharmacodynamic profile of THC oral formulations with Dronabinol as comparator
- THC F3 (Experimental): Drug: THC:CBC Oral solution of THC (5 mg/mL) & CBC (5 mg/mL)
  Interventions: Drug: Pharmacokinetic and pharmacodynamic profile of THC oral formulations with Dronabinol as comparator

INTERVENTIONS:
Drug: Pharmacokinetic and pharmacodynamic profile of THC oral formulations with Dronabinol as comparator — Assessment of Pharmacokinetic and pharmacodynamic profile of THC oral formulations in 4 arms in healthy volunteers and patients post-chemotherapy.
  Other Names: Administration of different Cannabis oral formulations with THC as compared with Active comparator (DRONABINOL)

SUMMARY:
Study based on the pharmacokinetic, pharmacodynamic, safety and stability evaluation of 3 standardized formulations of THC, to be used in healthy volunteers and post-chemotherapy patients as an adjuvant in the symptomatic treatment of the latter in discomfort associated with cancer treatment, with the aim of possible new therapeutic entities.

DETAILED DESCRIPTION:
This evaluation project of 3 oral formulations of Δ9-THC will be carried out in two phases: Phase I evaluation of bioequivalences in healthy subjects and Phase II evaluation of safety and effectiveness comparing with the reference product (Dronabinol 5mg/mL), formulations derived from cannabis for the management of nausea, vomiting post chemotherapy and exploratory in cancer pain.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy volunteers

In order to be eligible to be admitted to this study, healthy volunteers must:

1. Being a person > 18 years of age
2. Have the ability to understand the requirements of the study and be willing to give written informed consent
3. Agree to abide by study restrictions and return for required evaluations.
4. Signed written informed consent.

Inclusion criteria for patients

In order to be eligible to be admitted to this study, patients must:

1. Being a person > 18 years of age
2. Be a patient with documented chemotherapy treatment.
3. Patients with any of the following cancers: breast, prostate, lung, colorectal, cervical, gastric and liver cancer.
4. Have a life expectancy >1 year
5. Have the ability to understand the requirements of the study and be willing to give written informed consent
6. Agree to abide by study restrictions and return for required evaluations

Exclusion Criteria:

Exclusion criteria for healthy volunteers

To be eligible to be admitted to this study, the participant and/or patient must not:

1. Recreational or medicinal use of cannabinoids in the last 3 months.
2. Uses of current medications such as: immunomodulators, antibiotics, corticosteroids
3. Hypersensitivity to any component of the investigational product.
4. Patients prescribed dronabinol between arrival and prior to screening/randomization
5. Pregnancy or lactation
6. Liver pathologies and/or CYP2A3, CYP2C9 and CYP2C19 polymorphisms
7. Opioid hypersensitivity
8. Obesity
9. Patients who have undergone concomitant immunotherapy with chemotherapy
10. Cannabinoid Hyperemesis Syndrome (CHS).

Exclusion criteria for patients

To be eligible to be admitted to this study, the participant and/or patient must not:

1. Patients who are null by mouth (NPO) at the time of randomization or who are expected to be NPO within the next 48 hours
2. Patients who have received or are expected to receive neuraxial/locoregional blocks for pain in the next 48 hours.
3. Recreational or medicinal use of cannabinoids in the last 3 months.
4. Uses of current medications such as: immunomodulators, antibiotics, corticosteroids
5. Hypersensitivity to any component of the investigational product.
6. Patients prescribed dronabinol between arrival and prior to screening/randomization
7. Pregnancy or lactation
8. Liver pathologies and/or CYP2A3, CYP2C9 and CYP2C19 polymorphisms
9. Opioid hypersensitivity
10. Obesity
11. Patients who have undergone concomitant immunotherapy with chemotherapy
12. Cannabinoid Hyperemesis Syndrome (CHS). -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic assessment profile of THC formulations | 48 hours with a replicate 7 days after the first dose in healthy subjects and the same time but with successive doses in post-chemotherapy patients
  Pharmacokinetics of THC by Assessment of Area Under the Curve From Time Zero Extrapolated to Infinity (AUC(0-inf)) [ Time Frame: 0 hours (pre-dose), as well as at 0.12, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose ]
Pharmacodynamic assessment profile of THC formulations: BPI | Post-chemotherapy patients for at least 20 days with a daily report
  Brief pain inventory (BPI); The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning. The questions ask participants to rate their pain in the prior 24-hours OR prior 7-day on a 0 to 10 Numerical Rating Scale (NRS), where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine."
Pharmacodynamic assessment profile of THC formulations: DEQ | 48 hours with a replicate of 7 days after the first dose in healthy subjects and on the other hand post-chemotherapy patients for at least 20 days with a daily report
  Drug Effects Questionnaire (DEQ);is used in studies of acute subjective response (SR) to a variety of substances. The DEQ consists of 11 questions: "Feel Drug", "Feel High", "Like Drug", and "Want More", "dislike the sensation", "any sensations", "feel a head rush", "like drug effect", "dislike any effects". To calculate the DEQ- 'Good Drug Effects'. Each question was measured on a scale with a minimum score of 0 and a maximum score of 100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome
No significant nausea in terms of the proportion of subjects with no significant nausea | Post-chemotherapy patients for at least 20 days with a daily report
  To investigate THC oral formulations in terms of the proportion of patients with no significant nausea (none or mild nausea) following initiation of oral formulations of THC (dronabinol) in post-chemotherapy patients

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 14 days for healthy subjects, 20 days for post-chemotherapy patients
  Evaluate the Safety and Tolerability of Oral Formulations of THC, Number of AEs during 14 days for healthy subjects and 20 days for post-chemotherapy patients vs active drug phase vs. Dronabinol active comparator
Global Quality of Life (QoL) of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire | at least 20 days for post-chemotherapy patients
  EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  Self-reported symptoms related to treatment. Each item is rated on a response scale 1 = not at all to 4 = very much and refer to the time frame "during the last days" EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Lasanta S A S, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided